CLINICAL TRIAL: NCT03820570
Title: Comparison of Early and Long Term Outcomes of Open Lichtenstein Repair and Totally Extraperitoneal Herniorrhaphy for Primary Inguinal Hernias
Brief Title: Comparison Open Lichtenstein Repair and Totally Extraperitoneal Herniorrhaphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEPP
Record Dates: First submitted 2018-10-23; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lichtenstein (Experimental): hernia repair
  Interventions: Procedure: hernia repair

INTERVENTIONS:
Procedure: hernia repair — inguinal hernia repair

SUMMARY:
comparison of early and long term results of open lichtenstein repair and totally extraperitoneal herniorrhaphy for primary inguinal hernias.

DETAILED DESCRIPTION:
Early results such as postoperative pain, operation time and long term results such as chronic pain and recurrence will be compared.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia

Exclusion Criteria:

* recurrent hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
recurrence | 3 years
  hernia recurrence